CLINICAL TRIAL: NCT05911750
Title: Prevalence and Clinical Implications of Human Papillomavirus Infection in the Male Population With Inflammatory Bowel Disease
Brief Title: Prevalence and Clinical Implications of HPV Infection in Male IBD Patients
Acronym: PAPIMALE
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-VHP-2023-47
Record Dates: First submitted 2023-05-30; First posted 2023-06-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-06

CONDITIONS: HPV Infection; Dysplasia Anus; Oral Cavity Disease
Keywords: HPV, oral swab, anal swab
MeSH Terms: conditions — Papillomavirus Infections; Mouth Diseases | interventions — Cytological Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Rectal and oral mucosal cells collected by anal and oral swab, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male IBD patients: Male patients with a confirmed diagnosis of Inflammatory Bowel Disease (Crohn´s disease or Ulcerative colitis).
  Interventions: Diagnostic Test: Anal pap smear and oral swab for cytology and HPV testing

INTERVENTIONS:
Diagnostic Test: Anal pap smear and oral swab for cytology and HPV testing — Anal and oral swab sampling for HPV detection (polymerase chain reaction) and cytology

SUMMARY:
The study aims at describing the prevalence of Human Papillomavirus (HPV) infection in anal and oral samples of men with Inflammatory Bowel Disease (IBD) and detecting risk factors for the infection.

DETAILED DESCRIPTION:
Male IBD patients attending the IBD Clinic of Hospital de la Santa Creu i Sant Pau will be screened for eligibility. Informed consent will be obtained from all eligible patients. An anal and oral swab will be performed on all patients to look for HPV infection (HPV DNA test) and cytologic alterations. Patients will be inspected to rule out the presence of HPV-related lesions. Moreover, a self-administered questionnaire will be completed by all enrolled patients. Information regarding IBD characteristics and treatment will be obtained.

According to local practice, patients with anal or oral squamous intraepithelial lesions (ASIL) will be referred to a colorectal surgeon for further recommendations or treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Crohn's disease or ulcerative colitis (at least 3 months before enrollment)
* Male
* Age from 18 to 79 years

Exclusion Criteria:

* Unclassified Inflammatory Bowel Disease
* Diarrhea (> 3 bowel movements/day) with rectal bleeding at enrollment
* Prior full proctectomy
* Inability to collect the biological samples
* Inability to complete the questionnaire
* Refusal to sign the informed consent

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male IBD patients referring to the IBD Clinic of Hospital de la Santa Creu i Sant Pau
Sampling Method: Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2023-02-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence (number/percentage) of HPV infection in oral and anal samples | Up to 12 months
  PCR analysis will identify the presence of HPV in oral or anal mucosal cells and characterize the genotype of HPV.
Prevalence (number/percentage) of abnormal HPV-related cytology in oral and anal samples | Up to 12 months
  Cytology changes will be reported according to the Bethesda classification.

SECONDARY OUTCOMES:
Multivariate analysis to identify risk factors for HPV infection in oral and anal samples. | Up to 12 months
  Risk factors such as demographics, sexual conduct, and factors related to Inflammatory Bowel Disease (IBD) and IBD therapy will be evaluated through patient history research and the use of a self-administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Giordano, MD, Principal Investigator — dr.antoniogiordano@gmail.com
Locations (1):
- Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
IPD will be only shared upon request and with IEC approval.